CLINICAL TRIAL: NCT00838929
Title: Phase I Study of the Combination of Vorinostat and Radiation Therapy for the Treatment of Patients With Brain Metastases
Brief Title: Study of the Combination of Vorinostat and Radiation Therapy for the Treatment of Patients With Brain Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08D.522; 2008-19 (Other: CCRRC); JT 1331 (Other: JeffTrial Number)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Brain Metastases
Keywords: brain metastases; radiation; vorinostat; lung cancer; breast cancer
MeSH Terms: conditions — Brain Neoplasms; Lung Neoplasms; Breast Neoplasms | interventions — Vorinostat; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vorinostat (200 mg) and radiation (Experimental): Cohort 1: Patients receive 200 mg of Vorinostat and radiation
  Interventions: Drug: Vorinostat; Radiation: Radiation Therapy
- Vorinostat (300 mg) and radiation (Experimental): Cohort 2: Patients receive 300 mg of vorinostat and radiation
  Interventions: Drug: Vorinostat; Radiation: Radiation Therapy
- Vorinostat (400 mg) and radiation (Experimental): Cohort 3: Patients receive 400 mg of vorinostat and radiation
  Interventions: Drug: Vorinostat; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Vorinostat — All doses given for 3 weeks
  Dose level -2 - 50 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level -1 - 100 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level I - 200 mg PO qd (initial starting dose) Dose level II - 300 mg PO qd Dose level III - 400 mg PO qd
  Other Names: Zolinza
Radiation: Radiation Therapy — Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
  Other Names: Radiation oncology; Radiotherapy; XRT

SUMMARY:
Vorinostat in combination with radiation therapy can be administered safely and will be tolerated in patients with brain metastases, while providing an assessment of the anti-tumor activity of this combination.

This is a multi-center, open-label, non-randomized Phase I study in patients with brain metastases. Patients will be administered oral Vorinostat and radiation therapy and will be treated for 3 weeks. Patients will be enrolled in cohorts and will be treated at sequentially rising dose levels of Vorinostat combined with radiation therapy. We will initially enter 3 subjects at each dose. If none of the three experiences a dose-limiting toxicity we will proceed to the next dose. If one of the three experiences that level of toxicity, we will accrue 3 more subjects at that dose. If at any time there are two or more dose-limiting toxicities (in the 3-6 subjects) on a given dose, we will drop down to a lower dose. Dose escalation will continue until the MTD of Vorinostat and radiation therapy is established. The MTD will then be one dose below the DLT occurring in at least 1 out of 3 subjects (2 out of 6 patients).

DETAILED DESCRIPTION:
In recent years, a number of investigators have shown that combining signal transduction agents with ionizing radiation results in significant antitumor effects without an increase in normal tissue toxicity. There are numerous lines of evidence that Histone deacetylase (HDAC) inhibitors have been shown to enhance the radiosensitivity of tumor cells in vitro and in vivo 1-6. Vorinostat (Zolinza, suberoylanilide hydroxamic acid - SAHA) a potent histone deacetylase, has recently been approved for clinical use for cutaneous T-cell lymphoma. It has the potential to inhibit tumor growth and proliferation7-13, tumor angiogenesis14 and enhance radiation response15 with minimal toxicity. This phase I study, is based on the range of efficacy of Vorinostat and its ability to cross the blood-brain barrier. This study will evaluate the safety of combination of Vorinostat and daily-fractionated radiation therapy. This information is critical for any combined future combined modality trials that involves radiation therapy to the brain.

Vorinostat was approved by the US Food and Drug Administration (FDA) on 6-Oct-2006 for the treatment of cutaneous manifestations in patients with cutaneous T-cell lymphoma (CTCL) who have progressive, persistent or recurrent disease on or following two systemic therapies.

Based on preclinical, clinical efficacy and safety data, it is anticipated that Vorinostat in combination with radiation therapy can be administered safely and will be tolerated in patients with brain metastases. In addition, within the recognized limits of a Phase I clinical trial, this study may provide an assessment of the anti-tumor activity of Vorinostat in combination with radiation therapy in patients with brain metastases.

The present study will investigate the safety, tolerability and spectrum of side effects of Vorinostat in combination with radiation therapy. As such, this study will characterize the dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of in combination with radiation therapy in patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring a 3 week course of fractionated whole brain radiation therapy for brain metastases.
2. Age > or = 18
3. Histological or cytological diagnosis of a malignancy.
4. Patients who have only 1-3 metastases are frequently treated with stereotactic radiation. Nonetheless, if the treating physician decides that whole brain radiotherapy is the appropriate treatment such patients would be eligible to enroll upon in the study.
5. Radiographic evidence of brain metastasis.
6. Measurable disease preferred but not required for eligibility
7. Patient must have performance status of < or = 2 on the ECOG Performance Scale.
8. Life expectancy of > or = 3 months
9. Resolution of all acute toxic effects of prior chemotherapy or radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade < or = 1.
10. Adequate organ function as defined by the following criteria:

    * Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) < or = 2.5 x local laboratory upper limit of normal (ULN), or AST and ALT < or = 5 x ULN if liver function abnormalities are due to underlying malignancy
    * Total serum bilirubin < or = 1.5 x ULN
    * Absolute neutrophil count (ANC) > or = 1500/µL
    * Platelets > or = 100,000/µL
    * Hemoglobin > or = 9.0 g/dL
    * Serum calcium < or = 12.0 mg/dL
    * Serum creatinine < or = 1.5 x ULN
    * Potassium level within normal limits.
    * Magnesium level within normal limits.
11. Female patient of childbearing potential has a negative serum pregnancy test β-hCG within 72 hours prior to receiving the first dose of Vorinostat .
12. Female patient is either post menopausal, free from menses for > or = 2 years, surgically sterilized, or willing to use 2 adequate barrier methods of contraception to prevent pregnancy, starting with Visit 1.
13. Male patient agrees to use an adequate method of contraception for the duration of the study.
14. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
15. INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of Vorinostat and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
16. Patient is available for study related assessments, and management at the treating institution, for the duration of the study.

Exclusion Criteria:

1. Previous cranial irradiation (whether whole or partial brain, single fraction or multiple fractions) within the previous six months.
2. Patient who has had chemotherapy within 21 days, non-cranial radiotherapy within 10 days, or who has not recovered from adverse events due to agents administered more than 30 days earlier.
3. Patient is currently participating or has participated in a study with an investigational compound or device within 14 days of initial dosing with study drug(s).
4. Patient has had prior treatment with an HDAC inhibitor (e.g., romidepsin (Depsipeptide), NSC-630176, MS 275, LAQ-824, belinostat (PXD-101), LBH589, MGCD0103, CRA024781, etc). Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period under neurological supervision.
5. Patients with markedly elevated intracranial pressure.
6. Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
7. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
8. An extended QTc interval on baseline EKG examination. Normal values: male < 430ms, female <450 ms.
9. Concomitant use of medications known to extend the QTc interval: Quinidine, Procainamide, Disopyramide, Dofetilide, Ibutilide, Sotalol, Amiodarone, Bepridil, Cisapride, Macrolides, Erythromycin, Clarithromycin, Fluoroquinolones, Sparfloxacin, Antiprotozoals, Pentamidine, Antimalarials, Halofantrine, Chloroquine, Phenothiazine neuroleptics, Thioridazine, Chlorpromazine, Mesoridazine, Butyrophenone neuroleptics, Droperidol, Haloperidol, Diphenylpiperidine neuroleptics, Pimozide, Arsenic trioxide, Methadone, Cesium, Licorice, Zhigancao
10. Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
11. Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
12. Active clinically serious infection > CTCAE Grade 2
13. NCI CTCAE grade 3 hemorrhage within 4 weeks of starting the study treatment.
14. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
15. Pulmonary hemorrhage/bleeding event > or = CTCAE Grade 2 within 4 weeks of first dose of study drug.
16. Serious non-healing wound, ulcer, or bone fracture.
17. Evidence or history of bleeding diathesis or coagulopathy
18. Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
19. Use of St. John's Wort or rifampin (rifampicin).
20. Any condition that impairs patient's ability to swallow whole pills.
21. Any malabsorption problem.
22. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
23. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
24. Documented history of cranial hemorrhage
25. Patient has an active infection or has received intravenous antibiotics, antiviral, or antifungal agents within 2 weeks prior to the start of the study drug.
26. Patient has uncontrolled inter-current illness or circumstances that could limit compliance with the study, including, but not limited to the following: active infection, acute or chronic graft versus host disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric conditions.
27. Patient has a history or current evidence of any condition, therapy, or lab abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study or is not in the best interest of the patient to participate.
28. Patient has a history of a gastrointestinal surgery or other procedures that might, in the opinion of the investigator, interfere with the absorption or swallowing of the study drugs.
29. Patient has known hypersensitivity to the components of study drug or its analogs.
30. Patient has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
31. Patient is, at the time of signing informed consent, a regular user (including "recreational use") of any illicit drugs, substance abuse or had a recent history (within the last year) of drug or alcohol abuse.
32. Patient is pregnant or breast feeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-03; Primary Completion 2012-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Thomas Jefferson Universtiy
Locations (2):
- United States (2):
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Vorinostat (200 mg) and Radiation: Patients will be treated on a dose escalation model for vorinostat and concurrently receive radiation therapy.
  Vorinostat : All doses given for 3 weeks
  Dose level -2 - 50 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level -1 - 100 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level I - 200 mg PO qd (initial starting dose) Dose level II - 300 mg PO qd Dose level III - 400 mg PO qd
  Radiation Therapy : Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
Period: Overall Study
Arm/Group | Vorinostat (200 mg) and Radiation | Vorinostat (300 mg) and Radiation | Vorinostat (400 mg) and Radiation
Started | 3 | 8 | 6
Completed | 3 | 5 | 5
Not Completed | 0 | 3 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Disease progression | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat (200 mg) and Radiation: Patients will be treated on a dose escalation model for vorinostat and concurrently receive radiation therapy.
  Vorinostat : All doses given for 3 weeks
  Dose level I - 200 mg PO qd (initial starting dose)
  Radiation Therapy : Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
- Vorinostat (300 mg) and Radiation: Patients will be treated on a dose escalation model for vorinostat and concurrently receive radiation therapy.
  Vorinostat : All doses given for 3 weeks
  Dose level II - 300 mg PO qd
  Radiation Therapy : Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
- Vorinostat (400 mg) and Radiation: Patients will be treated on a dose escalation model for vorinostat and concurrently receive radiation therapy.
  Vorinostat : All doses given for 3 weeks
  Dose level III - 400 mg PO qd
  Radiation Therapy : Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
- Total: Total of all reporting groups
Arm/Group | Vorinostat (200 mg) and Radiation | Vorinostat (300 mg) and Radiation | Vorinostat (400 mg) and Radiation | Total
Number analyzed (Participants) | 3 | 8 | 6 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 5 | 10
  >=65 years | 3 | 3 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 9
  Male | 2 | 3 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 8 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of Vorinostat and Radiotherapy in Patients With Brain Metastases.
Description: To determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of Vorinostat and radiotherapy in patients with brain metastases.
  The maximum tolerated dose (MTD) will be one dose below the DLT occurring in at least 1 out of 3 subjects.
  Dose level -2: 50 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level -1: 100 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level I: 200 mg PO qd (initial starting dose) Dose level II: 300 mg PO qd Dose level III: 400 mg PO qd
Time Frame: Weekly during treatment On Last day of treatment (30 days after last drug dose) Follow-up (every 3 months)
Measure: Number; unit: mg
Groups:
- Vorinostat and Radiation - All Participants: Patients will be treated on a dose escalation model for vorinostat and concurrently receive radiation therapy.
  Vorinostat : All doses given for 3 weeks
  Dose level -2 - 50 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level -1 - 100 mg PO qd (to be used in de-escalation if toxicity occurs) Dose level I - 200 mg PO qd (initial starting dose) Dose level II - 300 mg PO qd Dose level III - 400 mg PO qd
  Radiation Therapy : Patients will take Vorinostat daily during radiation therapy, they will be recommended to swallow the capsule 60-90 minutes prior to estimate time of radiation.
Arm/Group | Vorinostat and Radiation - All Participants
Number analyzed (Participants) | 13
mg | 300

ADVERSE EVENTS:
Arm/Group | Vorinostat (200 mg) and Radiation | Vorinostat (300 mg) and Radiation | Vorinostat (400 mg) and Radiation
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 3/6
Other Adverse Events (participants affected / at risk) | 2/3 | 6/7 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (200 mg) and Radiation (N=3) | Vorinostat (300 mg) and Radiation (N=7) | Vorinostat (400 mg) and Radiation (N=6)
Increase in amylase (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) — Disease progession
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ulceration - Grade 3 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (200 mg) and Radiation (N=3) | Vorinostat (300 mg) and Radiation (N=7) | Vorinostat (400 mg) and Radiation (N=6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oral pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Ulceration - Grade 2 (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (General disorders) | 0 (0) | 1 (1) | 1 (1)
Partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Increased blood alkaline phosphatase (General disorders) | 0 (0) | 1 (1) | 0 (0)
Low hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Increased alanine aminotransferase (General disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Low platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Low sodium (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes